CLINICAL TRIAL: NCT05496985
Title: Chinese Validation of the Simplified Evaluation of CONsciousness Disorders（SECONDs）
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Haibo Di, professor, Hangzhou Normal University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: YCYY-20211021-003
Record Dates: First submitted 2022-08-01; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Brain Diseases; Vegetative State; Unconsciousness; Central Nervous System Diseases
Keywords: coma; disorder of consciousness; behavioral scale; rehabilitation; diagnosis
MeSH Terms: conditions — Brain Diseases; Persistent Vegetative State; Unconsciousness; Central Nervous System Diseases; Coma; Consciousness Disorders; Disease

STUDY DESIGN:
Intervention Model Description: Each patient was assessed by three distinct assessors who were experienced and trained to use the CRS-R. All assessments were completed within two weeks (i.e., five CRS-R to obtain a reliable diagnosis [17], and 7 SECONDs performed by 3 different assessors in the 2 weeks) in five different sessions. Session 1 included one evaluation with the CRS-R performed by one assessor (i.e., concurrent validity) and three evaluations with the SECONDs performed by two assessors (i.e., intra-rater reliability and inter-rater reliability). The other sessions (2 to 5) each included one evaluation with the SECONDs and one evaluation with the CRS-R (i.e., concurrent validity) performed by two assessors. Each SECONDs was performed alternatively either before or after the CRS-R assessment. To avoid fatigue effects and reduce the impact of within-day fluctuations of vigilance, a break of 30 to 80 min between each assessment was taken.
Who Masked: Outcomes Assessor
Masking Description: Until the end of the protocol, all three assessors were blinded to the scores acquired by the other assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients in coma (Experimental): Patients in coma were assessed by the SECONDs and CRS-R for five days.
  Interventions: Diagnostic Test: Simplified Evaluation of CONsciousness Disorders (SECONDs)
- Patients in unresponsive wakefulness syndrome (Experimental): Patients in unresponsive wakefulness syndrome were assessed by the SECONDs and CRS-R for five days.
  Interventions: Diagnostic Test: Simplified Evaluation of CONsciousness Disorders (SECONDs)
- Patients in minimally conscious state (Experimental): Patients in minimally conscious state were assessed by the SECONDs and CRS-R for five days.
  Interventions: Diagnostic Test: Simplified Evaluation of CONsciousness Disorders (SECONDs)
- Patients in emerge from the minimally conscious state (Experimental): Patients in emerge from the minimally conscious state were assessed by the SECONDs and CRS-R for five days.
  Interventions: Diagnostic Test: Simplified Evaluation of CONsciousness Disorders (SECONDs)

INTERVENTIONS:
Diagnostic Test: Simplified Evaluation of CONsciousness Disorders (SECONDs) — All patients were assessed by the Simplified Evaluation of CONsciousness Disorders (SECONDs) and Coma Recovery Scale-Revised (CRS-R)

SUMMARY:
The aim of this study was to translate the SECONDs from French into Chinese and assess the validity and reliability of the Chinese version of the SECONDs .

DETAILED DESCRIPTION:
To promote accurate assessments of DoC patients and the development of clinical research on DoC in China, we here propose and validate a version of the SECONDs translated into Mandarin Chinese. Hence, this study aims to assess the concurrent validity (compared with the CRS-R which has already been translated and validated in Mandarin), intra-rater reliability, and inter-rater reliability of the Chinese version of the SECONDs

ELIGIBILITY:
Inclusion Criteria:

* Acute (longer than 14 days, less than 28 days) or prolonged DoC (following severe acquired brain injury, longer than 28 days);
* Age: 18-85 years old;
* No history of other neurological or psychiatric deficits;
* Ability to speak Chinese fluently;
* Medical stability (e.g., absence of mechanical ventilation, sedation, infection)

Exclusion Criteria:

* None

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Assess the reliability and validity of the Chinese version of the SECONDs | Within 10 days
  The reliability and validity of the Chinese version of the SECONDs were evaluated by calculating the weighted Cohen's Kappa and Spearman coefficients of the differences between SECONDs and CRS-R in the diagnosis of MCS and UWS patients
Diagnose the level of consciousness in patients through SECONDs and CRS-R | Within 10 days
  Detect acute (longer than 14 days, less than 28 days) or prolonged DoC (following severe acquired brain injury, longer than 28 days) patients through Simplified Evaluation of CONsciousness Disorders (SECONDs).
Diagnose the level of consciousness in patients through CRS-R | Within 10 days
  Detect acute (longer than 14 days, less than 28 days) or prolonged DoC (following severe acquired brain injury, longer than 28 days) patients through Coma Recovery Scale-Revised (CRS-R).

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Di, Study Director — International Vegetative State and Consciousness Science Institute,Hangzhou Normal University; Anqi Wang, Principal Investigator — International Vegetative State and Consciousness Science Institute,Hangzhou Normal University
Locations (1):
- International Vegetative State and Consciousness Science Institute, Hangzhou Normal University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No